CLINICAL TRIAL: NCT05755945
Title: A Prospective Feasibility Study Evaluating the Use of Wearable Devices to Predict and Track Clinical Outcomes in Chronic Migraine
Brief Title: A Study of Wearable Devices to Predict Migraines
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Narayan R. Kissoon, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-009944
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Custom Phone eHealth Application (Experimental): Subjects diagnosed with migraine headaches and have had a positive response to prevention treatments for migraine, will wear an Apple Watch whenever possible (including during sleep) and complete application questionnaires on the eHealth application daily.
  Interventions: Other: eHealth Application

INTERVENTIONS:
Other: eHealth Application — Custom phone application that integrates data from smart watch. Subjects will complete daily "To-Do-Lists" where data will be collected on if they had a headache in the past 24 hours, severity of headache, and any analgesics used to treat the headache.

SUMMARY:
The purpose of this research is to determine if data from smart devices, including heart rate and movement during sleep and wake times, will be able to track headaches and predict recurrence and exacerbations (make worse). This use of this information may in the future allow patients earlier and more effective treatments if these devices can help predict when the headaches may occur.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older (no upper age limit defined)
* History of chronic migraine as defined by the International Headache Society's International Classification of Headache Disorders (3rd edition).
* Response to current preventative therapy with ≥ 50% improvement in the frequency of headache days when compared to baseline
* 4 to 14 average number of total headache days per month during peak efficacy of preventative therapy
* Ability to understand study procedures and to comply with them for the entire length of the study and use study devices as outlined in protocol.
* Patient agrees to maintain a daily electronic headache diary.
* Proficient in the use of electronic devices including Apple HomeKit and Apple Watch. - Subjects owns an iPhone with iOS 16 or later operating system installed on iPhone. Apple watch series 8 with watch OS6 or later will be provided by the study.

Exclusion Criteria:

* Chronic daily headache with no periods of headache freedom.
* ≥ 15 average number of headaches days per month during peak efficacy of preventative treatment.
* Medication overuse headache as defined by the International Headache Society's International Classification of Headache Disorders (3rd edition).
* Daily opioid use for > 3 months (e.g., hydrocodone, oxycodone, fentanyl patch) or other daily analgesic use for chronic pain disorders (e.g., NSAIDS or acetaminophen).
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage accuracy of fit with AUC of the ROC (receiver operating characteristics) curve (%) for headache tracking. | 6 months
  Percentage accuracy of fit with AUC of the ROC curve for factors from data collected from custom phone app integrated with smart devices to track headache frequency and severity.

SECONDARY OUTCOMES:
Percentage accuracy of fit with AUC of the ROC curve (%) for headache forecasting. | 6 months
  Percentage accuracy of fit with AUC of the ROC curve for data from custom phone app integrated with smart devices to forecast periods of increased headache likelihood.
Correlation coefficients of wearable sensor data to headache frequency and severity. | 6 months
  Correlation of novel physiological clinical outcome data (e.g., time in bed, average sleep time, stand time, exercise time, move time, walking distance, running distance, estimated six-minute walk, steps per day, heart rate, heart rate variability) to monthly headache days, moderate to severe monthly headache days, analgesic use, MIDAS, and HIT-6.
uMARS app quality mean score | 6 months
  Quality of the custom phone app integrated with smart watches as assessed by the validated uMARS.

CONTACTS AND LOCATIONS:
Overall Officials: Naraya Kissoon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials